CLINICAL TRIAL: NCT06401278
Title: Trans Cutaneous Electrical Acupoint Stimulation Versus TENS On Blood Pressure And Quality Of Life In Patients With Primary Hypertension
Brief Title: Trans Cutaneous Electrical Acupoint Stimulation Versus TENS On Blood Pressure In Primary Hypertension Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tawfik Tawfik Mahmoud Emara (Other)
Responsible Party: Sponsor-Investigator, Tawfik Tawfik Mahmoud Emara, Assistant Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004443
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Quality of Life
MeSH Terms: conditions — Hypertension | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous electrical acupoint stimulation (Group A): (Experimental): Transcutaneous electrical acupoint stimulation :It will be performed by using the TENS device on acupoint (TEAS) as the following:
  The patients will be placed in a relaxed comfortable sitting position with their back well supported. for 40 min three times weekly for a total of 6 weeks.The adhesive electrodes of the TENS device will be placed on the selected acupoint bilaterally Nei-Guan (PC6), Taichong (LR3), and Sanyinjiao (SP6)
  Interventions: Device: Transcutaneous electrical acupoint stimulation
- Transcutaneous electrical nerve stimulation(Group b): (Experimental): TENS will be applied in the cervicothoracic ganglion region located between the C7 and T4 vertebral processes for 40 min three times weekly for a total of 6 weeks.
  Interventions: Device: Transcutaneous electrical nerve stimulation (group b):
- Control (No Intervention): Routine medical treatment: (Group c): receive only routine medical treatment (antihypertensive medication, instructions and education to control blood pressure)
  * Nutrition Eat a diet that is high in fiber and potassium, and low in salt (sodium), added sugar, and fat.
  * Lifestyle Do not use any products that contain nicotine or tobacco, such as cigarettes, and chewing tobacco.
  * Identify your sources of stress and find ways to manage stress. This may include deep breathing or making time for fun activities.
  * Do not drink alcohol

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — It will be performed by using the TENS device on acupoint (TEAS) as the following:
  The patients will be placed in a relaxed comfortable sitting position with their back well supported. for 40 min three times weekly for a total of 6 weeks.The adhesive electrodes of the TENS device will be placed on the selected acupoint bilaterally Nei-Guan (PC6), Taichong (LR3), and Sanyinjiao (SP6)
  Arms: Transcutaneous electrical acupoint stimulation (Group A):
Device: Transcutaneous electrical nerve stimulation (group b): — TENS will be applied in the cervicothoracic ganglion region located between the C7 and T4 vertebral processes for 40 min three times weekly for a total of 6 weeks.
  Arms: Transcutaneous electrical nerve stimulation(Group b):

SUMMARY:
To compare between the effects of transcutaneous electrical acupoint stimulation and TENS on blood pressure and quality of life in patients with primary hypertension

BACKGROUND:

The current American College of Cardiology and the American Heart Association (ACC/AHA) 2017 guidelines define hypertension as systolic BP (SBP) of ≥130 mmHg or diastolic BP (DBP) of ≥80 mmHg. In adults, an increase of 20 mmHg in SBP or 10 mmHg in DBP is associated with more than a two-fold increase in mortality owing to stroke and other cardiovascular diseases. Hypertension accounts for 13% of premature deaths worldwide and is the third leading cause of disability-adjusted life years (Shah et al., 2022).

Transcutaneous electrical nerve stimulation of the Neiguan (P6) point with acupressure is possibly affecting the blood pressure by protecting the myocardial tissues and influencing the nervous system through regulating the autonomic nervous system function and reduction in sympathetic activity. (Hassanein et al., 2021).

HYPOTHESES There will be no a significant difference between the effects of transcutaneous electrical acupoint stimulation and TENS on blood pressure and quality of life in patients with primary hypertension

RESEARCH QUESTION:

Is there a significant difference between the effects of transcutaneous electrical acupoint stimulation and TENS on blood pressure and quality of life in patients with primary hypertension?

Evaluating equipment, pre-post intervension outcomes:

1. BP by Digital Sphygmomanometer
2. quality of life by The SF-12 health status questionnaire
3. nitric oxide level in blood by nitric Oxide analysis.
4. sleep quality. by Pittsburgh Sleep Quality Index (PSQI)
5. exercise capacity and endurance by Thirty-Second Sit-To-Stand Test (30 STST)

ELIGIBILITY:
Inclusion Criteria:

* 1) Sixty patients from both sexes diagnosed with essential HT at least 6 months ago.

  2) Their age will be ranged from 50 to 60 years old. 3) Their blood pressure will be ranged from (SBP is 140 -159 mmHg and/or DBP is 90-99 mmHg).

  4) Their body mass index (BMI) ranged from will be ranged from 24.9 to 29.9 kg/m2.

  5) All patients are medically stable and receive the same medical treatment 6) All patient nonsmoker or quitted smoking for at least 4-5 years 7) All patients will be similar in terms of status of functional activity, status of eating a salt-free diet and the presence of any chronic disease except HT

Exclusion Criteria:

* 1) Secondary hypertension 2) Patients with cardiac problems e.g. atrial fibrillation, left bundle-branch block, heart failure, recent myocardial infarction, coronary artery disease, or participation in cardiac rehabilitation following bypass surgery.

  3) Patients with history, symptoms of, and/or laboratory reports suggestive of renal, neurologic, or hepatic complications.

  4) Use of a cardiac pacemaker 5) Any metal implants at site of application of TENS 6) Dermatological abnormalities at the site of the application of TENS 7) Obesity with body mass index (BMI) > 30 kg/m2 8) Smoker, diabetes. 9) Soft tissue, nerve, and vascular diseases of upper or lower extremities which hinder the application of TEAS.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-08-05 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure by using a digital sphygmomanometer | six weeks
  Blood pressure was recorded by using a digital sphygmomanometer
quality of life by Short Form twelve health status questionnaire | six weeks
  by Short Form twelve health status questionnaire Health-Related Quality of Life survey consisting of twelve questions that measure eight health domains to assess physical and mental health.The score ranges from 0 to 100, with a higher score indicating better physical and mental health functioning.
Nitric oxide by nitric oxide sample analysis | six weeks
  by nitric oxide sample analysis

SECONDARY OUTCOMES:
exercise capacity and endurance measured by Thirty-Second Sit-To-Stand Test (30 STST) | six weeks
  measured by Thirty-Second Sit-To-Stand Test (30 STST)
sleep quality | six weeks
  Measured by Pittsburgh Sleep Quality Index (PSQI) It assesses sleep quality through seven components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction) which the participant is asked to recall over the past month. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality than lowest component.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy- Cairo Uni., Giza, Egypt

IPD SHARING:
Plan to Share IPD: No